CLINICAL TRIAL: NCT04767048
Title: Interest of Bilateral Basic Tongue Mucosectomy Assisted by Robot or Laser in Combination with Tonsillectomy in the Assessment of Prevalent Cervical Lymphadenopathy: a Randomized Phase II Study
Brief Title: Interest of Bilateral Basic Tongue Mucosectomy Assisted by Robot or Laser in Combination with Tonsillectomy in the Assessment of Prevalent Cervical Lymphadenopathy
Acronym: RoboCUP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A00947-32
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cancer of Head and Neck; Adenopathy
Keywords: mucosectomy; tonsil
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphadenopathy | interventions — Tonsillectomy

STUDY DESIGN:
Masking Description: tonsillectomy +/- bilateral mucosectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Basic bilateral tongue mucosectomy assisted by robot or laser plus tonsillectomy (unilateral or bilateral at the choice of the investigator)
  Interventions: Procedure: bilateral mucosectomy + tonsillectomy
- Control Arm (Active Comparator): Tonsillectomy alone (unilateral or bilateral at the choice of the investigator)
  Interventions: Procedure: tonsillectomy

INTERVENTIONS:
Procedure: bilateral mucosectomy + tonsillectomy — Basic bilateral tongue mucosectomy assisted by robot or laser plus tonsillectomy (unilateral or bilateral at the choice of the investigator)
  Arms: Experimental Arm
Procedure: tonsillectomy — tonsillectomy (unilateral or bilateral at the choice of the investigator)
  Arms: Control Arm

SUMMARY:
We are proposing a randomized phase II study to assess the benefit of bilateral robot-assisted or laser basal tongue mucosectomy in combination with tonsillectomy in the assessment of prevalent cervical lymphadenopathy

ELIGIBILITY:
Inclusion Criteria:

* Patient with a prevalent head and neck lymphadenopathy with positive or non-contributory fine needle aspiration, or having had an adenectomy revealing a metastasis of squamous cell carcinoma, a PET examination, an injected cervico-thoracic CT and an ENT work-up (nasofibroscopy) not finding a primary tumor
* Performance Status < 2
* Patient aged 18 or over
* Patient affiliated with social security system
* Informed consent signed

Exclusion Criteria:

* History of squamous cell carcinoma of the VADS or skin of the face.
* History of cervico-facial radiotherapy
* Primary tumor discovering during pan-endoscopy
* Inexposable patient lead not to possible mucosectomy
* Uncontrollable hemostasis disorders (contraindication to tonsillectomy and basic bilateral mucosectomy of language)
* Distant metastases
* Lymphadenopathy inoperable
* Patient with a contraindication to radiotherapy
* Pregnant or breastfeeding woman
* Women of childbearing potential without effective contraception
* Patient under guardianship or unable to give informed consent
* Patient unable to undergo the trial follow-up for geographic, social or psychopathological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Detection of primary cancer | At surgery
  Proportion of patients with primary cancer detected with surgery

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre François Baclesse, Caen
  - CHU CAEN, Caen
  - Centre Oscar Lambret, Lille
  - Chru Lille, Lille
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bastit V, Lequesne J, Leconte A, Deneuve S, Mouawad F, Quak E, Jeanne C, Clarisse B, Thariat J. Effectiveness of bilateral tongue base mucosectomy by transoral robotic surgery or transoral laser microsurgery in combination with tonsillectomy in identifying head and neck primary cancer of unknown primary: a randomized phase 2 protocol (RoboCUP trial). BMC Cancer. 2025 Mar 27;25(1):551. doi: 10.1186/s12885-025-13913-7. PMID 40148848